CLINICAL TRIAL: NCT06502990
Title: Open-label, Phase 3b Study to Evaluate Effectiveness, Safety and Pharmacokinetic Parameters of Metreleptin in Patients Under 6 Years of Age With Generalised Lipodystrophy and Associated Diabetes Mellitus and/or Hypertriglyceridaemia
Brief Title: Open-label Study to Evaluate Metreleptin in Children Under 6 Years of Age With Generalised Lipodystrophy
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Amryt Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APL-20; 2022-501781-22-00 (EU CTIS Number)
Record Dates: First submitted 2024-07-09; First posted 2024-07-16 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Generalized Lipodystrophy
Keywords: Metreleptin
MeSH Terms: conditions — Lipodystrophy, Congenital Generalized | interventions — metreleptin

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Metreleptin (Experimental): Metreleptin [Recombinant-methionyl human Leptin; rmetHuLeptin] for daily injection is a sterile, white, solid lyophilised cake
  Interventions: Drug: Metreleptin

INTERVENTIONS:
Drug: Metreleptin — Metreleptin is a recombinant human leptin analog that is indicated as an adjunct to diet as replacement therapy to treat the complications of leptin deficiency

SUMMARY:
This is an open-label, Phase 3b study to evaluate effectiveness, safety and pharmacokinetic parameters of metreleptin in patients under 6 years of age with generalised lipodystrophy and associated diabetes mellitus and/or hypertriglyceridaemia

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of Generalised Lipodystrophy
* Metreleptin treatment naive

Exclusion Criteria:

* Weight <9 kg at Screening (Visit 1)

Max Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Estimated)
Dates: Start 2025-05-23 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Percent change from baseline in fasting serum TG levels at Month 12 for subjects with fasting TG levels ≥2.3 mmol/L (200 mg/dL) at baseline | 12 months
  To evaluate the effectiveness of metreleptin in patients under 6 years of age with GL and associated diabetes mellitus and/or hypertriglyceridaemia
Absolute change from baseline in glycated haemoglobin (HbA1c) at Month 12 for subjects with HbA1c ≥6.5% at baseline | 12 months
  To evaluate the effectiveness of metreleptin in patients under 6 years of age with GL and associated diabetes mellitus and/or hypertriglyceridaemia

SECONDARY OUTCOMES:
Proportion of subjects of those with Baseline HbA1c ≥6.5% achieving target actual decreases of at least 0.5%, 1%, 1.5%, 2% absolute decrease in HbA1c or HbA1c <6.5% or HbA1c <5.7% at Month 12 | 12 months
  To evaluate the efficacy of metreleptin treatment in patients with GL
Proportion of subjects of those with Baseline HbA1c ≥5.7% achieving target actual decreases of at least 0.5%, 1%, 1.5%, 2% absolute decrease in HbA1c or HbA1c <5.7% at Month 12 | 12 months
  To evaluate the efficacy of metreleptin treatment in patients with GL
Proportion of subjects of those with fasting serum TG ≥ 1.7 mmol/L (150 mg/dL) achieving target actual decreases from baseline of at least 15%, 20%, 25%, 30%, 35%, 40% at Month 12 | 12 months
  To evaluate the efficacy of metreleptin treatment in patients with GL
Proportion of subjects of those with fasting serum TG ≥ 2.3 mmol/L (200 mg/dL) achieving target actual decreases from baseline of at least 15%, 20%, 25%, 30%, 35%, 40% at Month 12 | 12 months
  To evaluate the efficacy of metreleptin treatment in patients with GL
Change from baseline in liver volume and liver span as assessed by ultrasound at each post-baseline visit through Month 12 | 12 months
  To evaluate the efficacy of metreleptin treatment in patients with GL
Incidence of, treatment emergent adverse events (TEAEs), serious adverse events (SAEs), treatment related adverse events (AEs), AEs of special interest (AESIs) and AEs leading to study drug discontinuation | 12 months
  To assess safety and tolerability of metreleptin

CONTACTS AND LOCATIONS:
Locations (12):
- UZ Leuven, Leuven, Belgium
- France (2):
  - Hôpital Necker - Enfants Malades, Paris
  - Assistance Publique-Hopitaux de Paris (AP-HP) - Hopital Universitaire Robert-Debre, Paris
- Germany (2):
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Universitaetsklinikum Ulm - Klinik fuer Kinder- und Jugendmedizin, Ulm
- Italy (7):
  - IRCCS Ospedale Pediatrico Bambino Gesù, Chieti
  - Azienda Ospedaliera Universitaria "Federico II", Naples
  - Azienda Ospedaliero Universitaria Maggiore della Carità di Novara, Novara
  - Azienda Ospedaliero-Universitaria di Parma, Parma
  - Azienda Ospedaliero Universitaria Pisana, Pisa
  - IRCCS Ospedale Pediatrico Bambino Gesù, Rome
  - Ospedale Filippo Del Ponte Varese - ASST Sette Laghi, Varese